CLINICAL TRIAL: NCT01350895
Title: Clinical and Biochemical Presentation of Polycystic Ovary Syndrome in Different Age Group
Status: Completed | Type: Observational
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Principal Investigator, Ming-I Hsu, Attending Doctor, Taipei Medical University WanFang Hospital
Other Study IDs: WFH-PCOS-100002
Record Dates: First submitted 2011-05-09; First posted 2011-05-10 (Estimated); Last update posted 2013-11-06 (Estimated); Status verified 2013-11

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Polycystic ovarian syndrome (PCOS)
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Experimental Group
- Control Group

SUMMARY:
To study the clinical and biochemical characteristics women with polycystic ovary syndrome (PCOS) in different aged groups.

DETAILED DESCRIPTION:
Polycystic ovarian syndrome (PCOS) is the most frequent endocrine disorder of reproductive age women, affecting an estimated 9-18% of all women in this age group. To diagnose of PCOS in early life is especially important because it is now thought to increase metabolic and cardiovascular risks. Investigating PCOS is crucial as it is now considered to increase metabolic and cardiovascular risk, thereby impacting the health of women to a much greater extent than previously thought. We are plan using retrospective analysis to evaluate the clinical and biochemical presentation of PCOS in different aged groups.

ELIGIBILITY:
Inclusion Criteria:

* Reproductive age women with sufficient data

Exclusion Criteria:

* Disorders of uterus (e.g. Asherman's Syndrome, Mullerian agenesis) and chromosomal anomalies (e.g. Turner syndrome)
* women who had had menarche at less than 3 years of age, Day 3 FSH > 15, or who were older than 46
* women with inadequate clinical/biochemical records
* and women who had had ovarian cysts or ovarian tumors in ultrasonography examination
* pregnancy women

Ages: 18 Years to 46 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Reproductive age women
Sampling Method: Non-Probability Sample
Enrollment: 781 (Actual)
Dates: Start 2011-02; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ming-I Hsu, Principal Investigator — Taipei Medical University WanFang Hospital
Locations (1):
- Taipei Medical University-WanFang Hospital, Taipei, Taiwan